CLINICAL TRIAL: NCT03827369
Title: The Blood Pressure Analysis on Critically Ill Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taoyuan General Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: TYGH107041
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Multiple Organ Failure; Intensive Care Unit Syndrome
Keywords: Blood pressure; Arterial pulse; Coefficient of variation of harmonic magnitude
MeSH Terms: conditions — Multiple Organ Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU patient: Pulse pressure of the radical artery was obtained by arterial line. The output of the transducer was connected to an IBM PC for analysis via an A/D converter with sampling rate = 250 datapoints/sec. The pulse spectrum was analyzed with the Fourier transformation using T (period) = 1 pulse time.
  Interventions: Diagnostic Test: ICU patient

INTERVENTIONS:
Diagnostic Test: ICU patient — Our study is to measure the coefficient of variation of the HCV of the radial arterial pulse among ICU patients with multiple organ failures (MOF). Patients admitted to Taoyuan General Hospital were recorded during the 6 months study.

SUMMARY:
The study is to explore the relationship between coefficient of variation of harmonic magnitude (HCV) and different organ failures among those critically ill patients. In the future, we can act as a warning system on patients with multiple organ failures or terminal illness, also as an indicator of treatment effect.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients in the 20-to-99 age range
* Subjects agree to sign the Informed Consent Form and are willing to cooperate with Arterial pulse measurement

Exclusion Criteria:

* Subject has severe arrhythmia

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients without severe arrhythmia admitted to the ICU of Taoyuan General Hospital.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-04-30 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Coefficient of variation of harmonic magnitude | 15 min
  We measure the blood pressure of participants with multiple organ failures (MOF) by pressure transducer during the 6 months study in the ICU of Taoyuan General Hospital. The radial artery pressure pulse of both hands are recorded with a pressure transducer fixed on the skin with tape and an adjustable belt with a small button to achieve suitable pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Tzu-Yi Chuang, Principal Investigator — Taoyuan General Hospital, Minstry of Healthy and Welfare
Locations (1):
- Taoyuan General Hospital, Ministry of Health and Welfare, Taoyuan District, Taiwan